CLINICAL TRIAL: NCT00417170
Title: A Double-blind, Double Dummy, Randomized Parallel Design Trial to Study the Effects of 12 Weeks of Treatment With 300mg Aliskiren vs. 5mg Amlodipine on Insulin Resistance and Endothelial Dysfunction in Hypertensive Patients With Metabolic Syndrome
Brief Title: Comparison of Aliskiren and Amlodipine on Insulin Resistance and Endothelial Dysfunction in Patients With Hypertension and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100A2239
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: High Blood Pressure; Metabolic Syndrome; Insulin Resistance; Endothelial Dysfunction
Keywords: High Blood pressure; Hypertension; metabolic syndrome; insulin resistance; endothelial dysfunction; pre-diabetic; amlodipine,; aliskiren,; IGT,; IFG,; MBF
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Insulin Resistance; Glucose Intolerance | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren 300 mg (Experimental): Eligible participants received oral Aliskiren 300 mg + Placebo Amlodipine once daily for 12 weeks. Study medication was taken with 200 mL of water in the morning. Breakfast was eaten 1 hour after taking study medication. Study medication was swallowed whole, and not chewed.
  Interventions: Drug: Aliskiren; Drug: Placebo Amlodipine
- Amlodipine 5 mg (Active Comparator): Eligible participants received oral Amlodipine 5 mg + Placebo Aliskiren once daily for 12 weeks. Study medication was taken with 200 mL of water in the morning. Breakfast was eaten 1 hour after taking study medication. Study medication was swallowed whole, and not chewed.
  Interventions: Drug: Amlodipine; Drug: Placebo Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg tablets taken orally once daily
  Arms: Aliskiren 300 mg
Drug: Amlodipine — Amlodipine 5 mg capsule taken orally once daily
  Arms: Amlodipine 5 mg
Drug: Placebo Aliskiren — Placebo Aliskiren taken orally once daily.
  Arms: Amlodipine 5 mg
Drug: Placebo Amlodipine — Placebo Amlodipine taken orally once daily
  Arms: Aliskiren 300 mg

SUMMARY:
The purpose of this study was to determine the effects of Aliskiren on insulin resistance (IR) and endothelial dysfunction (ED) in patients with high blood pressure and metabolic syndrome. The efficacy of Aliskiren was compared to Amlodipine.

ELIGIBILITY:
Inclusion criteria:

* Male or female adults aged 18 to 55 years, inclusive.
* Sitting diastolic blood pressure ≥80 mm Hg and/or sitting systolic blood pressure ≥ 130 at screening.
* Metabolic Syndrome as defined by the Adult Treatment Panel (ATP) III criteria.
* Hypertension (defined above) and impaired glucose tolerance (IGT) or impaired fasting glucose (IFG) plus one or more out of the remaining 3 criteria to satisfy entry into the study. IGT and IFG will be classified according to American Diabetes Association (ADA) guidelines:

  * IFG: Fasting plasma glucose of 100 mg/dl (5.6 mmol/l) to 125 mg/dl (6.9 mmol/l)
  * IGT: Two-hour plasma glucose of 140 mg/dl (7.8 mmol/l) to 199 mg/dl (11.0 mmol/l)
* Abnormal Positron Emission Tomography (PET) results at baseline. (Myocardial Blood Flow (MBF) of less than or equal to 35%.)
* Abnormal euglycemic clamp results at baseline. (Glucose infusion rate (GINF) of less than or equal to 4.2 mg/kg/min.)
* Body mass index (BMI) of less than 40.

Exclusion criteria:

* Smokers (use of tobacco products in the recent past)
* Cardiovascular abnormalities including myocardial infarction, angina pectoris, hypertensive encephalopathy, stroke, transient ischemic attack, valvular heart disease, ventricular arrhythmia, A-V block, atrial fibrillation or cardiac revascularization/angioplasty in the past 12 months.
* Symptoms or clinical evidence of congestive heart failure or known left ventricular ejection fraction < 40%.
* Supine Blood pressure ≥ 160 mmHg systolic or ≥110 mmHg diastolic.
* Clinically significant echocardiogram (ECG) abnormalities, including history of a prolonged QT-interval syndrome.
* Significant autonomic dysfunction.
* Severe bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* Clinically significant drug allergy, atopic allergy (asthma, urticaria, eczematous dermatitis).
* Pregnant or breastfeeding females. Pre-menopausal females who are not practicing a non-hormonal method of birth control.
* African Americans will not be eligible for this study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Santa Monica, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening for eligibility took place up to 6 weeks prior to study start. Participants stopped taking all medications during the 6 week screening period and washed out of all medications, including antihypertensive medication prior to randomization and start of study dosing.
Groups:
- Aliskiren 300 mg: Aliskiren 300 mg + Placebo Amlodipine orally once daily for 12 weeks.
- Amlodipine 5 mg: Amlodipine 5 mg + Placebo Aliskiren orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Started | 23 ("Started" indicates Safety population.) | 25
Pharmacodynamics Population | 21 | 23
Completed | 21 | 22
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg | Total
Number analyzed (Participants) | 23 | 25 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11.3) | 44.1 (5.3) | 44.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 7 | 17 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Endothelial Function as Measured by Myocardial Blood Flow (MBF) From Baseline and After 12 Weeks of Treatment
Description: MBF is measured by Positron Emission Tomography (PET) first at rest, then 45 minutes later, during cold pressor testing (CPT). The patient is placed in the PET scanner and injected with N-13 ammonia as a tracer. PET images are taken to assess myocardial blood flow at rest. After 40 minutes, the patient immerses one hand in ice water and PET images are taken to assess myocardial blood flow at sympathetic activation. Change from baseline data is analyzed by an analysis of variance (ANOVA) model including treatment and week as fixed factors and subject (nested in treatment) as a random factor.
Time Frame: At baseline and after 12 weeks of treatment
Population: The Pharmacodynamic (PD) analysis set includes all participants with available PD data and no major protocol deviation with impact on PD data. Participants with observations at both baseline and endpoint were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mL/g/min
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Number analyzed (Participants) | 21 | 23
mL/g/min | 0.06 (0.39) | 0.12 (0.39)

2. Secondary Outcome: Mean Change in Insulin Sensitivity as Measured by Glucose Infusion Rate (Last 30 Minutes) From Baseline and After 12 Weeks of Treatment.
Description: Insulin sensitivity is measured by the hyperglycemic euglycemic clamp procedure where a supine patient has 2 IV lines inserted for sampling blood. Regular human insulin (60mU/m^2 surface area/min) is infused for 120 minutes. Dextrose (20% w/v) is infused to maintain glycemia at < 100 mg/dL and is adjusted based on plasma glucose levels obtained every 5 minutes. Blood for glucose and insulin is taken at specified time intervals. Change from baseline data is analyzed by analysis of variance model including treatment and week as fixed factors, and subject (nested in treatment) as a random factor.
Time Frame: At baseline and after 12 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/kg/min
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Number analyzed (Participants) | 21 | 22
mg/kg/min | 0.23 (0.379) | 0.55 (0.371)

3. Secondary Outcome: Mean Change in Insulin Concentration as Measured During Oral Glucose Tolerance Test (OGTT) From Baseline and After 12 Weeks of Treatment
Description: Insulin Concentration is determined by the Oral Glucose Tolerance Test (OGTT) which begins after a 10 hour overnight fast. Blood samples are taken at baseline and after an oral 75 gram dose of glucose. Additional samples of blood are taken to measure glucose and insulin levels at 30, 60, 120 and 180 minutes post glucose intake. Changes from pre-glucose intake values are analyzed by an analysis of variance (ANOVA) model including treatment, visit and post-dose time points ( 30, 60, 120 and 180 minutes) as fixed factors and subject (nested in treatment) as a random factor.
Time Frame: At baseline and after 12 weeks of treatment
Population: The Pharmacodynamic (PD) analysis set included all participants with available PD data and no major protocol deviation with impact on PD data. During different time points, participants with observations at that time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mU/L
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Number analyzed (Participants) | 21 | 23
mU/L
  0 minutes (n=21, 23) | 3.54 (14.666) | -3.08 (14.014)
  30 minutes (n=17, 21) | 31.26 (15.748) | -15.46 (14.436)
  60 minutes (n=19, 22) | 16.71 (15.169) | -27.87 (14.231)
  120 minutes (n=17, 19) | 33.27 (15.745) | -52.67 (14.930)
  180 minutes (n=19, 22) | 22.96 (15.144) | -43.58 (14.231)

4. Secondary Outcome: Mean Change From Baseline in Inflammatory Marker ( C-peptide) as Measured During Oral Glucose Tolerance Test (OGTT) From Baseline and After 12 Weeks of Treatment [Time Frame: At Baseline and After 12 Weeks of Treatment
Description: C-peptide level is determined by the Oral Glucose Tolerance Test (OGTT) which begins after a 10 hour overnight fast. Blood samples are taken at baseline and after an oral 75 gram dose of glucose. Additional samples of blood are taken to measure glucose and insulin levels at 30, 60, 120 and 180 minutes post glucose intake. Changes from pre-glucose intake values are analyzed by an analysis of variance (ANOVA) model including treatment, visit and post-dose time points ( 30, 60, 120 and 180 minutes) as fixed factors and subject (nested in treatment) as a random factor.
Time Frame: Baseline and after 12 weeks of treatment
Population: The PD analysis set included all subjects with available PD data and no major protocol deviations with impact on PD data. During different time points, participants with observations at that time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Number analyzed (Participants) | 21 | 23
ng/mL
  0 minutes ( n = 21, 23) | 0.302 (0.3891) | -0.215 (0.3718)
  30 minutes ( n= 20, 22) | 0.862 (0.3987) | -0.888 (0.3802)

5. Secondary Outcome: Mean Change in Arterial Compliance as Measured by Pulse Wave Analysis From Baseline and After 12 Weeks of Treatment
Description: Arterial Compliance is determined by Pulse Wave Analysis measured by a detector placed at the carotid artery while taking ECG and tonometry at the same time. Procedure is repeated for the femoral artery. Pulse Wave data are calculated by dividing distance between 2 arteries by the difference between the rise delay of the distal pulse wave and the R wave of the QRS complex and the rise delay of the proximal pulse wave to the QRS complex. Data analysis used an analysis of variance (ANOVA) model including treatment and week as fixed factors and subject (nested in treatment) as a random factor.
Time Frame: At baseline and after 12 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren 300 mg | Amlodipine 5 mg
Number analyzed (Participants) | 20 | 21
mmHg
  Central Systolic Blood Pressure | -17.7 (2.22) [upper limit NA] | -11.1 (2.19) [NA to NA]
  Central Mean Pressure | -1.39 (0.158) [NA to NA] | -0.85 (0.156) [NA to NA]
  Central Diastolic Blood Pressure | -11.0 (1.38) [NA to NA] | -6.3 (1.36) [NA to NA]
  Systolic Blood Pressure (Peripheral) | -16.2 (2.15) [NA to NA] | -10.0 (2.12) [NA to NA]
  Diastolic Blood Pressure (Peripheral) | -10.6 (1.34) [NA to NA] | -6.0 (1.32) [NA to NA]

ADVERSE EVENTS:
Groups:
- Aliskiren 300mg: Aliskiren 300 mg + Placebo Amlodipine orally once daily for 12 weeks.
- Amlodipine 5mg: Amlodipine 5 mg + Placebo Aliskiren orally once daily for 12 weeks.
Arm/Group | Aliskiren 300mg | Amlodipine 5mg
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 2/23 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300mg (N=23) | Amlodipine 5mg (N=25)
OEDEMA PERIPHERAL (General disorders) | 0 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
GLUCOSE TOLERANCE INCREASED (Investigations) | 0 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.